CLINICAL TRIAL: NCT01403961
Title: Hemoglobin A1c and Immediate Postsurgical Complications Diabetes Type 2 (HbA1c)
Brief Title: Hemoglobin A1c and Immediate Postsurgical Complications Diabetes Type 2
Acronym: HbA1c
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Diego Hernan Giunta, MD, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 1439
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HbA1c > 7: Diabetic patients with HbA1c > 7
- HbA1c ≤ 7: Diabetic patients with HbA1c ≤ 7

SUMMARY:
The purpose of this study is to evaluate Hemoglobin A1c values previous to a surgery in patients with diabetes type II and the complication incidence in immediate post surgery.

DETAILED DESCRIPTION:
The diabetes is a highly prevalent disease in patients who undergo an evaluation previous to a surgery. The most efficient glucose control, in patients with diabetes type II, reduces the risk of microvascular complications. Diabectic patients who underwent scheduled cardivacular or noncardiovascular surgeries show an increase rate of immediate and long-term complications. The most frequent complications are infections, cardiovascular events and death.

Intensive insulinisation during cardiovascular surgery reduces the risk of a new coronary event in the immediate post surgery. No studies have been found that show the evaluation of Hemoglobin A1c values before the surgery and the immediate post surgery complications.

A poor glycemic control has been associated to a large number of chronic complications like diabetic neuropathy, nephropathy, retinopathy and infection disease. The Hemoglobin A1c is used like a marker of the glycemic control in the last 120 days and has a correlation with the no enzyme glicosilation. This marker could have a relation with the complication after the programmed surgery.

This study will evaluate the incidence of complications in the immediate post operatory in patients with diabetes type II in relation to the hemoglobin A1c before the surgery. If the hemoglobin A1c has a correlation with the incidence of cardiovascular complications, this could mark a change in the therapeutic measures prior the programmed surgery.

ELIGIBILITY:
Inclusion Criteria

1. Patients older than 18 years with diagnosed of diabetes type 2
2. Programmed major surgery with expected hospitalization longer than 24 hours

Exclusion Criteria

1. Refusal to participate in the study or the informed consent process.
2. Programmed cardiac or coronary surgery
3. Technical complications inherent to surgical or anatomical abnormalities.
4. Pregnant women.
5. Active infection prior to performing surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult diabetic patients
Sampling Method: Probability Sample
Enrollment: 1760 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Compare incidence of immediate post surgery complications in diabetic patients with HbA1c > 7 and patients with HbA1c ≤ 7 | 30 days postsurgery
  Incidence of death, infections, cardiovascular o brainvascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Diego Giunta, MD, Principal Investigator — AIMI. HIBA.; Javier GIunta, MD, Study Director — HIBA; Carlos Bonofiglio, MD, Study Chair — HIBA; Leon Litwak, MD, Study Chair — HIBA
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No